CLINICAL TRIAL: NCT05116722
Title: Shoulder Pacemaker for the Treatment of Scapular Dyskinesia
Brief Title: Shoulder Pacemaker for Scapular Dyskinesia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Tashjian, Principle Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 144053
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Scapular Dyskinesis; Posterior Shoulder Instability
Keywords: Scapular Dyskinesia; Posterior Shoulder Instability; Shoulder Pacemaker; Treatment; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Shoulder Pacemaker Treatment (Experimental): The patients will be treated using the pacemaker for 15 - 30 minutes at 3-months, 6-months and 12-months during physical therapy.
  Interventions: Device: Shoulder Pacemaker

INTERVENTIONS:
Device: Shoulder Pacemaker — Shoulder pacemaker treatment for 15 - 30 minutes at 3-months, 6-months and 12-months during physical therapy.

SUMMARY:
The investigators purpose of this study is to determine patients-reported outcomes (VAS pain scores) in patients with Scapular Dyskinesis or Posterior Shoulder Instability who undergo rehabilitation with a shoulder pacemaker.

DETAILED DESCRIPTION:
The scapula plays a key role in nearly every aspect of normal shoulder function. Shoulder dyskinesia or scapula winging effects patients as a result of nerve injury or muscle detachment or abnormal muscle recruitment. Patients with abnormal muscle recruitment often are helped the most by therapy but restoring normal firing can be difficult. Abnormal muscle recruitment is due to pain or weakness or instability of the glenohumeral joint and the muscles around the scapula attempt to compensate for the lack of normal firing patterns. In many patients, physical therapy and surgery have proven to be unsuccessful treatment options.

The Shoulder Pacemaker is a device that specifically aims at resolving functional issues that surgery and physical therapy are unable. It's a wearable electro stimulator created for patients suffering from unbalanced muscle activation in the shoulder, such as Scapular Dyskinesis. The Shoulder Pacemaker delivers "smart stimulation" through a dynamic interaction between the patient and the device. The motion technology recognizes muscle movement and automatically sets the appropriate stimulation intensity according to the movement. This process helps to restore normal muscle activation patterns and equilibrium. The pacemaker will hopefully assist in restoring normal muscle recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Scapular Dyskinesis
* Posterior Shoulder Instability

Exclusion Criteria:

* Rotator Cuff Tearing
* Shoulder Arthritis
* Patients with implantable electrical/electronic devices
* If participants are using wearable electrical medical devices, such as glucose sensors or infusion pumps, these devices will be turned off or the participants will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain | Beginning of the study prior to initiating use of the pacemaker
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 3-months
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 6-months
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 12-months
  VAS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Z Tashjian, MD, Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University Of Utah Orthopedics Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No